CLINICAL TRIAL: NCT04302012
Title: Assessment of EyeArt Performance With Retinal Imaging Devices
Status: Completed | Type: Observational
Sponsor: Eyenuk, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EN-01a
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Mydriatics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Procedure: Color fundus photography — Subjects will undergo fundus photography before and/or after administration of mydriatic agent
Drug: Mydriatic Agent — Subjects may be administered mydriatic medication to dilate their pupils.

SUMMARY:
The study evaluates the performance of the EyeArt system for detecting diabetic retinopathy from images captured using multiple retinal imaging devices and operators.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of diabetes mellitus;
* Understanding of study and provision of written informed consent; and
* 22 years of age or older.

Exclusion Criteria:

* Persistent visual impairment in one or both eyes;
* History of macular edema, severe non-proliferative retinopathy, proliferative retinopathy, or retinal vascular (vein or artery) occlusion;
* History of ocular injections, laser treatment of the retina, or intraocular surgery other than cataract surgery without complications;
* Subject is contraindicated for fundus photography (for example, has light sensitivity);
* Subject has contraindications for mydriatic medications or is unwilling or unable to dilate;
* Subject is currently enrolled in an interventional study of an investigational device or drug; or
* Subject has a condition or is in a situation which in the opinion of the Investigator, might confound study results, may interfere significantly with the subject's participation in the study, or may result in ungradable dilated fundus photographs.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects will be enrolled at primary care and/or eye care centers
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Agreement between multiple EyeArt operations | 1 visit (1 day)

CONTACTS AND LOCATIONS:
Locations (1):
- Lundquist Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No